CLINICAL TRIAL: NCT06860334
Title: UMIT-2: A Randomized, Multi-country, Adaptive Phase IIb Platform Trial to Determine the Efficacy and Safety of Therapeutics for Crimean-Congo Haemorrhagic Fever
Brief Title: UMIT-2 - Adaptive Phase IIb Platform Trial to Determine the Efficacy and Safety of Therapeutics for CCHF
Acronym: UMIT-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-013
Record Dates: First submitted 2025-02-13; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Crimean-Congo Hemorrhagic Fever
Keywords: CCHF; Favipiravir; Ribavirin; Crimean Congo Hemorrhagic Fever
MeSH Terms: conditions — Hemorrhagic Fever, Crimean | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomised open-label phase 2b trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimised standard of care (oSOC) (Active Comparator): Optimised standard of care will include treatment per national guidelines for CCHF case management in Turkiye and Iraq, and any other supportive medication or therapies as required. The standard of care arm will exclude any medicine defined as investigation arms of this study. Any supportive medication or therapies will be recorded on the patient CRFs.
  Interventions: Other: Optimised Standard of Care
- Arm B: Favipiravir (Active Comparator): Day 1 (First 24 hours): IV Favipiravir 2600 mg twice daily (BD) Day 2 (24-48 hours): IV Favipiravir 1200 mg twice daily (BD) Day 3 -7 (Post 48 hours): Oral (PO) Favipiravir 1200 mg twice daily (BD)1 until hospital discharge up to 7 days (14 doses) whichever is soonest.
  Plus any additional supportive care deemed necessary by the study investigator
  Interventions: Drug: Favipiravir
- Arm C: Ribavirin (Active Comparator): Day 1 (First 24 hours): IV Ribavirin (33mg/kg) loading dose followed by IV Ribavirin 16mg/kg every 6 hours Day 2 (24-48 hours): IV Ribavirin 16mg/kg four times daily (QDS) Days 3-5: Oral (PO) Ribavirin 16mg/kg four times daily (QDS) Days 6 -7: Oral (PO) Ribavirin 8mg/kg four times daily (QDS) until hospital discharge
  Plus any additional supportive care deemed necessary by the study investigator
  Interventions: Drug: Ribavin

INTERVENTIONS:
Drug: Favipiravir — 6-fluoro-3-hydroxypyrazine-2-carboxamide, T-705
  Arms: Arm B: Favipiravir
Drug: Ribavin — 1-3,4-dihydroxy-5-1,2,4-triazole-3-carboxamide
  Arms: Arm C: Ribavirin
Other: Optimised Standard of Care — Optimised standard of care will include treatment per national guidelines for CCHF case management in Turkiye and Iraq, and any other supportive medication or therapies as required.
  Arms: Optimised standard of care (oSOC)

SUMMARY:
CCHF has a wide geographical distribution with cases mainly occurring in Asia, the Middle East, South-Eastern Europe and Africa. Since its emergence in 2002, Turkiye has been the epicentre of activity worldwide reporting up to more than 1000 cases annually. CCHF case management relies on the provision of optimised supportive care; therapeutic options lack a robust evidence base

The UMIT-2 Trial (UMIT = 'Hope' in Turkish) will be the first large randomised controlled trial of novel therapeutics in CCHF, undertaken in multiple trial sites in Turkiye and Iraq. It uses an efficient adaptive platform design (Phase IIb), focussed on antiviral efficacy with interim monitoring to introduce new arms and allow early stopping for futility, efficacy, or safety

DETAILED DESCRIPTION:
This will be a 1:1:1 randomised open-label phase 2b trial of Favipiravir (IV & PO) and Ribavirin (IV & PO) vs optimised standard of care in CCHF aimed at evaluating virological efficacy. This is an adaptive multi-arm Phase II platform for patients with CCHF. Key design features are:

Treatment arms can be added or removed.

Shared standard of care (SoC, control) arm so that a greater proportion of more patients receive experimental therapeutics. Eligibility to randomisation to specific treatment arms is based on treatment specific inclusion/exclusion criteria and all comparisons to SoC are within the same eligibility set and concurrent randomisation.

Timing of interim analyses flexible to make use of the seasonality of CCHF to ensure they take place during low recruitment periods.

ELIGIBILITY:
Inclusion Criteria:

Adult in-patients (≥18 years)

Laboratory confirmed CCHF infection by positive polymerase chain reaction (PCR) test within 5 days prior to randomisation

Capacity to provide informed consent signed by study patient or legally acceptable representative (for illiterate individuals).

Women of childbearing potential (WOCBP) and male patients who are sexually active with WOCBP must agree to use a highly effective method of contraception (as outlined in section 5.4 below) from the first administration of trial treatment, throughout trial treatment and for the duration outlined in trial protocol as well as addition 14 days for women and 7 days for men after the last dose of trial treatment.

Severity Grading System (SGS) for CCHF - mild/moderate.

Less than or equal to 7 days from onset of CCHF symptoms

Willingness to participate in the full protocol

Requirement to be hospitalised for treatment-

Exclusion Criteria:

Stage 4 severe chronic kidney disease or requiring dialysis (i.e., estimated glomerular filtration (eGFR) rate <30 mL/min/1.73 m2)

Pregnant or breast feeding

Anticipated transfer to another hospital which is not a study site within 72 hours

Known Allergy to any study medication

Patients participating in another clinical trial of an investigational medicinal product (CTIMP) within the last 30 days.

Previous intolerance of Favipiravir or Ribavirin

Any participants deemed not suitable, based on investigators opinion.

Patients taking the drugs listed below within 30 days or 5 times the half-life (whichever is longer) of enrolment:

Pyrazinamide: Pyrazinamide administration with favipiravir examined possible renal urate transporter interactions. Pyrazinamide increased blood uric acid levels 2 to 9 mg/dL over baseline. The addition of favipiravir increased blood uric acid levels 4 to 11 mg/dL over baseline, indicating a moderate additive effect.

Repaglinide: Favipiravir administration with repaglinide, an anti-diabetic agent that is extensively metabolized by CYP2C8 and CYP3A4, increased repaglinide plasma AUC 30 to 50% due to inhibition of CYP2C8.

Theophylline: Theophylline administration with favipiravir increases plasma Cmax and AUC of favipiravir through xanthine oxidase (XO) interaction. The primary metabolite of theophylline is known to be metabolized by XO which is partially involved in metabolism of favipiravir.

Famciclovir, Sulindac: Famciclovir and Sulindac are converted to active metabolite by Aldehyde Oxidase (AO). Favipiravir inhibits AO and decrease the concentration of active metabolite of Famciclovir and Sulindac.

Paracetamol: Coadministration of paracetamol (650 mg once daily) and favipiravir (1200 mg twice daily or 800 mg twice daily) increased paracetamol Cmax and AUC by 3% and 16% (1200 mg doses) and by 8% and 14% (800 mg doses). In the UMIT-2 trial after screening and randomisation the daily dose of paracetamol in adults should be no more than 3000 mg/day (rather than 4000 mg/day) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Virologic objective: To compare CCHFV viral dynamics of investigational therapeutics relative to the control arm | Day 5 from treatment start
  Comparison of CCHFV viral load clearance by Day 5 for treatment arms compared to Standard of Care arm.

SECONDARY OUTCOMES:
Safety Objective: To determine the safety and tolerability of investigational therapeutics relative to the control arm | Day 29
  Comparison of incidence of serious adverse events in treatment arms compared to standard of care arm.
  Comparison of the frequency and characterisation of clinically significant adverse events related to study agent administration
  (Safety and Tolerability of Favipiravir and Ribavirin CTCAE v5 Grade ≥3 adverse events)
Clinical Objective: To compare time to successful hospital discharge between participants receiving investigational therapeutics, relative to the control arm | Day 29
  Time from Randomisation to discharge from hospital
Antiviral Objective: To evaluate antiviral efficacy of investigational therapeutics (1) | Day 10
  Comparison of CCHFV viral load reduction between for treatment arms compared to Standard of Care arm
Antiviral Objective: To evaluate antiviral efficacy of investigational therapeutics (2) | Day 10
  Comparison of Viral load reduction by PCR test for treatment arms compared to Standard of Care arm
Safety Objective: To compare the overall mortality in patients with CCHF who receive different investigational therapeutics with those who receive the control arm | Day 28
  Mortality at Days 14 and 28 (time from date of randomisation to death) for treatment arms compared to Standard of Care arm
Safety Objective: To compare mortality rates among patients whose baseline predictors of disease place them in different categories for disease severity, who receive different investigational therapeutics. | Day 28
  Mortality at Days 14 and 28 (time from date of randomisation to death) in different SGS groups for treatment arms compared to Standard of Care arm
Pharmacokinetic objective:To characterise the plasma pharmacokinetics (PK) of therapeutics in CCHF | Day 29
  To investigate the exposure-response relationship of Favipiravir on CCHF viral dynamics by analysing concentrations of investigation therapeutics in plasma

OTHER OUTCOMES:
To characterise virus, host immune response and viral resistance over time | Day 29
  Change in host immune response, CCHFV culture and sequencing related to study agent administration